CLINICAL TRIAL: NCT07390682
Title: Impact of Obesity on the Efficacy of Bilateral Tibial Nerve Stimulation in Obstructed Defecation
Brief Title: Obesity on the Efficacy of Bilateral Tibial Nerve Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Professor of General surgery, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: obesity and ODS
Record Dates: First submitted 2025-12-23; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Obstructed Defecation
Keywords: Obesity; Bilateral Tibial Nerve Stimulation; Obstructed Defecation; ODS; BT PTNS
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- obese with ODS (Active Comparator): BT PTNS in obese patients with ODS
  Interventions: Procedure: Bilateral posterior tibial nerve stimulation
- Non obese with ODS (Active Comparator): BT PTNS in non-obese patients with ODS
  Interventions: Procedure: Bilateral posterior tibial nerve stimulation

INTERVENTIONS:
Procedure: Bilateral posterior tibial nerve stimulation — * Procedure: BT PTNS will be administered via transcutaneous electrodes placed bilaterally along the posterior tibial nerve at the medial malleolus.
  * Frequency: 3 sessions per week for 6 weeks (total of 18 sessions).
  * Duration per Session: 30 minutes.
  * Monitoring: Patients will be monitored for adverse events during and after each session.

SUMMARY:
Obstructed defecation syndrome (ODS) is a common functional bowel disorder characterized by difficulty in stool evacuation. Bilateral posterior tibial nerve stimulation (BT PTNS) has emerged as a noninvasive, safe, and effective therapeutic option for functional ODS, improving symptom severity and quality of life.

DETAILED DESCRIPTION:
Obesity is associated with altered pelvic floor mechanics, which may affect the response to neuromodulation therapy. However, the effect of obesity on BT PTNS outcomes in ODS has not been systematically evaluated. This study aims to fill this knowledge gap by comparing treatment efficacy between obese and non-obese patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of functional obstructed defecation (Rome IV criteria).
* Able to provide informed consent.
* BMI ≥30 kg/m² (obese group) or BMI <30 kg/m² (non-obese group).

Exclusion Criteria:

* Organic causes of constipation (e.g., colorectal cancer, inflammatory bowel disease).
* Previous pelvic floor surgery.
* Neurological disorders affecting bowel function.
* Pregnancy or lactation.
* Current use of other neuromodulation therapies.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in symptom severity measured by the Modified Obstructed Defecation Score (MODS). | Within 6 weeks of treatment.
  Scale range: 0 to 24
  Interpretation: Higher scores indicate more severe obstructed defecation symptoms
  Unit of measure: Units on a validated symptom severity scale. No aggregation of different measurements into a single reported value is performed. Each scale is analyzed independently.
  In response to the Advisory Issue, we have included the unabbreviated titles of the scales, their minimum and maximum values, and clarified whether higher scores represent better or worse outcomes for each outcome measure.
Change in quality of life measured by the Patient Assessment of Constipation Quality of Life questionnaire (PAC-QOL). | Within 6 weeks of treatment.
  Scale range: 0 to 96
  Interpretation: Higher scores indicate worse constipation-related quality of life
  Unit of measure: Mean score on a validated quality-of-life scale No aggregation of different measurements into a single reported value is performed. Each scale is analyzed independently.
  In response to the Advisory Issue, we have included the unabbreviated titles of the scales, their minimum and maximum values, and clarified whether higher scores represent better or worse outcomes for each outcome measure.

SECONDARY OUTCOMES:
Pelvic floor function | Within 6 weeks of treatment.
  To assess the impact of obesity on pelvic floor function using electromyography (EMG).
  Electromyograpghy (EMG) a diagnostic test that evaluates the electrical signals between your nerves and muscles to check for neuromuscular problems like nerve damage or muscle diseases. It usually involves two parts: a nerve conduction study (NCS) using surface electrodes to measure nerve signal speed, and a needle EMG where a tiny needle electrode is inserted into a muscle to record its activity at rest and during contraction, revealing abnormalities. To assess amplitude, number of turns and duration of pelvic floor muscle.

CONTACTS AND LOCATIONS:
Locations (1):
- The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Undecided